CLINICAL TRIAL: NCT06399185
Title: Effect of Dexmedetomidine and Esketamine on Catheter-related Bladder Discomfort in Patients Undergoing Transurethral Surgery: a 2 x 2 Factorial Randomized Trial
Brief Title: Effect of Dexmedetomidine and Esketamine on Catheter-related Bladder Discomfort
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-105
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Urinary Catheter; Catheter-related Bladder Discomfort; Dexmedetomidine; Esketamine
Keywords: Urinary Catheter; Catheter-related Bladder Discomfort; Dexmedetomidine; Esketamine
MeSH Terms: interventions — Saline Solution; Dexmedetomidine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): 20 ml of normal saline is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Interventions: Drug: Normal saline
- Dexmedetomidine group (Experimental): Dexmedetomidine 0.5 μg/kg, diluted with normal saline to 20 ml, is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Interventions: Drug: Dexmedetomidine
- Esketamine group (Experimental): Esketamine 0.25 mg/kg, diluted with normal saline to 20 ml, is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Interventions: Drug: Esketamine
- Dexmedetomidine-esketamine group (Experimental): Dexmedetomidine 0.5 μg/kg and esketamine 0.25 mg/kg, diluted with normal saline to 20 ml, is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Interventions: Drug: Combined dexmedetomidine-esketamine

INTERVENTIONS:
Drug: Normal saline — 20 ml of normal saline is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Other Names: Placebo
  Arms: Placebo group
Drug: Dexmedetomidine — Dexmedetomidine 0.5 μg/kg, diluted with normal salinet o 20 ml, is infused intravenously at 60 ml/h after anesthesia induction but before surgery.
  Arms: Dexmedetomidine group
Drug: Esketamine — Esketamine 0.25 mg/kg, diluted with normal saline to 20 ml, is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Arms: Esketamine group
Drug: Combined dexmedetomidine-esketamine — Dexmedetomidine 0.5 μg/kg and esketamine 0.25 mg/kg, diluted with normal saline to 20 ml, is infused intravenously at 80 ml/h after anesthesia induction but before surgery.
  Arms: Dexmedetomidine-esketamine group

SUMMARY:
Catheter-related bladder discomfort (CRBD) is common in patients awaking from general anesthesia with an urinary catheter. We suppose that that use of dexmedetomidine and/or esketamine during anesthesia may reduce the occurrence of CRBD. This 2x2 factorial randomized trial is designed to explore the effects of esketamine, dexmedetomidine, and their combination on the occurrence CRBD in patients undergoing transurethral urological surgery.

DETAILED DESCRIPTION:
Urethral catheterization is commonly used during and after surgery. However, patients with indwelling urinary catheters often present with catheter-related bladder discomfort (CRBD) after awakening from anesthesia. CRBD is characterized by pain and discomfort in the suprapubic area or symptoms like overactive bladder, characterized by frequent and urgent urination, with or without acute incontinence. The incidence of CRBD is relatively high, ranging from 47% to 90%. The development of CRBD not only reduces patients' perioperative satisfaction, but also increases the incidence of postoperative complications, affects patients' postoperative rehabilitation, and prolongs the length of hospital stay. It also increases the workload of medical staff.

The occurrence of CRBD is affected by many factors, such as gender, size of urinary tube, and type of surgery. Studies show that the use of ≥18F catheter increases the incidence of CRBD. After transurethral surgery, such as transurethral resection of bladder tumor (TUR-Bt), transurethral resection of prostate (TURP), and transurethral holmium laser resection of prostate (HoLRP), a 20F catheter is often required for bladder irrigation; the catheter carrying time may be extended for bladder perfusion. Therefore, the incidence of CRBD is higher after such operations.

Dexmedetomidine is a highly selective α2 receptor agonist with analgesic, anxiolytic, and sedative effects. Several randomized trial confirmed that intraoperative use of 0.3-1.0 μg/kg dexmedetomidine reduces the incidence and severity of postoperative CRBD, and the effect persists up to 6 hours after surgery. Ketamine is a non-competitive N-methyl-D-aspartate receptor antagonist and produces analgesic and anti-hyperalgesia effects. A recent meta-analysis found that subanesthetic doses of ketamine (0.25 mg/kg or 0.5 mg/kg) reduce the severity of CRBD within 1-2 hours after surgery and the incidence of CRBD within 2-6 hours after surgery. Esketamine is the S-enantiomer of racemic ketamine and has a higher affinity for NMDA receptors; it is twice as potent as racemic ketamine.

The investigators hypothesize that the combination of dexmedetomidine and esketamine may improve the efficacy in preventing CRBD. This 2x2 factorial trial is designed to observe the effect of dexmedetomidine, esketamine, and dexmedetomidine-esketamine combination on the occurrence of CRBD in patients following transurethral urological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above;
* Scheduled to undergo transurethral bladder or prostate surgery (including transurethral resection of bladder tumor, transurethral resection of prostate, and transurethral thulium laser prostatectomy) under general anesthesia;
* Required postoperative retention of a three-chamber urinary catheter.

Exclusion Criteria:

* Indwelling urinary catheters or chronic analgesic therapy for ≥1 month before surgery;
* Uncontrolled hypertension before surgery (resting ward systolic pressure >180 mmHg or diastolic pressure >110 mmHg);
* Severe bradycardia (heart rate ≤50 beats per minute), sick sinus syndrome, or atrioventricular block of degree II or above without pacemaker, or having myocardial infarction, severe heart insufficiency (New York Heart Association class ≥3), or tachyarrhythmia within a year;
* Preoperative history of schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, or intracranial hypertension;
* Preoperative history of hyperthyroidism and pheochromocytoma;
* Inability to communicate due to coma, severe dementia, or language barrier before surgery;
* Severe liver dysfunction (Child-Pugh grade C), severe renal dysfunction (receiving dialysis before surgery), or Amercian Society of Anesthesiologists classification ≥IV;
* Scheduled admission to the intensive care unit with endotracheal intubation after surgery;
* Other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1740 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheter-related bladder discomfort (CRBD) within 24 hours after surgery. | Up to 24 hours after surgery.
  Defined as occurrence of moderate or severe CRBD at any time point within 24 hours after surgery. CRBD is a strong desire to urinate or discomfort in the pubic region that occurs after awakening from anesthesia. The occurrence of CRBD is assessed at 0 hour (arriving post-anesthesia care unit), 1 hour, 2 hours, 6 hours, and 24 hours after surgery. The severity of CRBD is divided into four levels: 1- None, even when asked, no discomfort is reported; 2- Mild, only report discomfort during questioning; 3-Moderate, reported discomfort without inquiry, but without behavioral reactions; 4-Severe, with the patient actively reporting discomfort and behavioral reactions (observable behavioral reactions include limb movement, strong vocal reactions, or attempts to remove the catheter).

SECONDARY OUTCOMES:
Prevalence of CRBD at various time points within 24 hours after surgery. | Up to 24 hours after surgery.
  The occurrence of CRBD is assessed at 0 hour (arriving post-anesthesia care unit), 1 hour, 2 hours, 6 hours, and 24 hours after surgery. The severity of CRBD is divided into four levels: 1- None, even when asked, no discomfort is reported; 2- Mild, only report discomfort during questioning; 3-Moderate, reported discomfort without inquiry, but without behavioral reactions; 4-Severe, with the patient actively reporting discomfort and behavioral reactions (observable behavioral reactions include limb movement, strong vocal reactions, or attempts to remove the catheter). A moderate or severe CRBD is defined as occurrence of CRBD.
Severity of CRBD at various time points within 24 hours after surgery. | Up to 24 hours after surgery.
  The occurrence of CRBD is assessed at 0 hour (arriving post-anesthesia care unit), 1 hour, 2 hours, 6 hours, and 24 hours after surgery. The severity of CRBD is divided into four levels: 1- None, even when asked, no discomfort is reported; 2- Mild, only report discomfort during questioning; 3-Moderate, reported discomfort without inquiry, but without behavioral reactions; 4-Severe, with the patient actively reporting discomfort and behavioral reactions (observable behavioral reactions include limb movement, strong vocal reactions, or attempts to remove the catheter).
Intensity of pain at various time points within 24 hours after surgery. | Up to 24 hours after surgery.
  Pain intensity both at rest and with movement is assessed with a numeric rating scale (an 11-point scale where 0=no pain and 10=the worst pain) at 0 hour (arriving post-anesthesia care unit), 1 hour, 2 hours, 6 hours, and 24 hours after surgery.
Subjective sleep quality on the night of surgery. | On the morning of the first postoperative day (8:00-10:00).
  Subjective sleep quality is assessed with a numeric rating scale (an 11-point scale where 0=the best sleep and 10=the worst sleep) on the morning of the first postoperative day (8:00-10:00).
Patient satisfaction at 6 hours after surgery. | At 6 hours after surgery.
  Patients' satisfaction with CRBD control is evaluated with a 7-point Likert scale: 1=very dissatisfied, 2=moderate dissatisfied, 3=mild dissatisfied, 4=no propensity (moderate), 5=mild satisfied, 6=moderate satisfied, 7=very satisfied.
Anxiety at hospital discharge or 2 days after surgery. | Up 2 days after surgery.
  Anxiety is assessed with Generalized Anxiety Disorder-7 (scores range from 0 to 21, with higher score indicating more severe anxiety).
Depression at hospital discharge or 2 days after surgery. | Up 2 days after surgery.
  Depression is assessed with Patient Health Questionnaire-9 (scores range from 0 to 27, with higher score indicating more severe depression.
Sleep quality at 30 days after surgery. | At 30 days after surgery.
  Sleep quality is assessed with the Pittsburgh Sleep Quality Index (PSQI) questionnaire, scores range from 0 to 21, with higher score indicating poorer sleep quality.

OTHER OUTCOMES:
Sedation or agitation score at various time points within 24 hours after surgery. | Up to 24 hours after surgery.
  Sedation or agitation score is assess with the Richmond Agitation-Sedation Scale (scores range from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm) at 0 hour (arriving post-anesthesia care unit), 1 hour, 2 hours, 6 hours, and 24 hours after surgery.
Use of rescue medications within 24 hours after surgery | Up to 24 hours after surgery.
  Rescue medications include opioids, non-steroid anti-inflammatory drugs, M-receptor blockers (totorodine, sorinaxin, mirabelon), and other analgesics for CRBD.
Duration of urinary catheterization after surgery. | Up to 30 days after surgery.
  Postoperative catheterization time
Length of hospital stay after surgery. | Up to 30 days after surgery.
  Length of hospital stay after surgery.
Occurrence of postoperative complications. | Up to 30 days after surgery.
  Postoperative complications are defined as newly occurred conditions that are deemed harmful to patients' recovery and required medical interventions, i.e., grade II or higher on Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson KE. Pharmacology of lower urinary tract smooth muscles and penile erectile tissues. Pharmacol Rev. 1993 Sep;45(3):253-308. No abstract available. PMID 8248281
- [Result] Binhas M, Motamed C, Hawajri N, Yiou R, Marty J. Predictors of catheter-related bladder discomfort in the post-anaesthesia care unit. Ann Fr Anesth Reanim. 2011 Feb;30(2):122-5. doi: 10.1016/j.annfar.2010.12.009. Epub 2011 Jan 31. PMID 21277735
- [Result] Bai Y, Wang X, Li X, Pu C, Yuan H, Tang Y, Li J, Wei Q, Han P. Management of Catheter-Related Bladder Discomfort in Patients Who Underwent Elective Surgery. J Endourol. 2015 Jun;29(6):640-9. doi: 10.1089/end.2014.0670. Epub 2014 Dec 9. PMID 25335575
- [Result] Mitobe Y, Yoshioka T, Baba Y, Yamaguchi Y, Nakagawa K, Itou T, Kurahashi K. Predictors of Catheter-Related Bladder Discomfort After Surgery: A Literature Review. J Clin Med Res. 2023 Apr;15(4):208-215. doi: 10.14740/jocmr4873. Epub 2023 Apr 28. PMID 37187710
- [Result] Moataz A, Chadli A, Wichou E, Gallouo M, Jandou I, Saber S, Serhier Z, Dakir M, Debbagh A, Aboutaieb R. [Predictors of catheter-related bladder discomfort]. Prog Urol. 2020 Dec;30(16):1045-1050. doi: 10.1016/j.purol.2020.09.014. Epub 2020 Sep 30. French. PMID 33011083
- [Result] Goger YE, Ozkent MS, Goger E, Kilinc MT, Ecer G, Piskin MM, Erol A. A randomised-controlled, prospective study on the effect of dorsal penile nerve block after TURP on catheter-related bladder discomfort and pain. Int J Clin Pract. 2021 May;75(5):e13963. doi: 10.1111/ijcp.13963. Epub 2021 Jan 11. PMID 33368991
- [Result] Wang SY, Qiu Q, Shen X. Effect of Pudendal Nerve Block on the Prevention of Postoperative Bladder Spasm and Catheter-Related Bladder Discomfort in Male Patients Undergoing Transurethral Holmium Laser Enucleation of the Prostate. Clin Interv Aging. 2022 Nov 30;17:1729-1738. doi: 10.2147/CIA.S384612. eCollection 2022. PMID 36474581
- [Result] Agarwal A, Yadav G, Gupta D, Singh PK, Singh U. Evaluation of intra-operative tramadol for prevention of catheter-related bladder discomfort: a prospective, randomized, double-blind study. Br J Anaesth. 2008 Oct;101(4):506-10. doi: 10.1093/bja/aen217. Epub 2008 Jul 24. PMID 18653496
- [Result] Zhang Z, Cao Z, Xu C, Wang H, Zhang C, Pan A, Wei R, Peng S, Guo F, Wang L, Sun Y. Solifenacin is able to improve the irritative symptoms after transurethral resection of bladder tumors. Urology. 2014 Jul;84(1):117-21. doi: 10.1016/j.urology.2014.02.034. Epub 2014 Apr 29. PMID 24785989
- [Result] Zhou Z, Cui Y, Zhang X, Lu Y, Chen Z, Zhang Y. The efficacy and safety of antimuscarinics for the prevention or treatment of catheter-related bladder discomfort: a systematic review and meta-analysis of randomized controlled trials. Perioper Med (Lond). 2021 Dec 14;10(1):46. doi: 10.1186/s13741-021-00217-0. PMID 34903279
- [Result] Li S, Li P, Wang R, Li H. Different interventions for preventing postoperative catheter-related bladder discomfort: a systematic review and meta-analysis. Eur J Clin Pharmacol. 2022 Jun;78(6):897-906. doi: 10.1007/s00228-021-03251-5. Epub 2022 Feb 26. PMID 35218404
- [Result] Ramesh R, Mittal A, Agrawal S. Pharmacological interventions for reducing catheter-related bladder discomfort in patients undergoing elective surgeries under general anaesthesia: A systematic review and meta-analysis. Indian J Anaesth. 2023 Feb;67(Suppl 2):S81-S92. doi: 10.4103/ija.ija_200_22. Epub 2023 Feb 22. PMID 37122936
- [Result] Srivastava VK, Nigam R, Agrawal S, Kumar S, Rambhad S, Kanaskar J. Evaluation of the efficacy of solifenacin and darifenacin for prevention of catheter-related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Minerva Anestesiol. 2016 Aug;82(8):867-73. PMID 27607187
- [Result] Agarwal A, Dhiraaj S, Singhal V, Kapoor R, Tandon M. Comparison of efficacy of oxybutynin and tolterodine for prevention of catheter related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Br J Anaesth. 2006 Mar;96(3):377-80. doi: 10.1093/bja/ael003. Epub 2006 Jan 16. PMID 16415311
- [Result] Fox C, Smith T, Maidment I, Chan WY, Bua N, Myint PK, Boustani M, Kwok CS, Glover M, Koopmans I, Campbell N. Effect of medications with anti-cholinergic properties on cognitive function, delirium, physical function and mortality: a systematic review. Age Ageing. 2014 Sep;43(5):604-15. doi: 10.1093/ageing/afu096. Epub 2014 Jul 19. PMID 25038833
- [Result] Oelke M, Speakman MJ, Desgrandchamps F, Mamoulakis C. Acute Urinary Retention Rates in the General Male Population and in Adult Men With Lower Urinary Tract Symptoms Participating in Pharmacotherapy Trials: A Literature Review. Urology. 2015 Oct;86(4):654-65. doi: 10.1016/j.urology.2015.06.025. Epub 2015 Jul 2. PMID 26142712
- [Result] Hur M, Park SK, Yoon HK, Yoo S, Lee HC, Kim WH, Kim JT, Ku JH, Bahk JH. Comparative effectiveness of interventions for managing postoperative catheter-related bladder discomfort: a systematic review and network meta-analysis. J Anesth. 2019 Apr;33(2):197-208. doi: 10.1007/s00540-018-2597-2. Epub 2019 Jan 2. PMID 30603826
- [Result] Takizuka A, Minami K, Uezono Y, Horishita T, Yokoyama T, Shiraishi M, Sakurai T, Shigematsu A, Ueta Y. Dexmedetomidine inhibits muscarinic type 3 receptors expressed in Xenopus oocytes and muscarine-induced intracellular Ca2+ elevation in cultured rat dorsal root ganglia cells. Naunyn Schmiedebergs Arch Pharmacol. 2007 Jul;375(5):293-301. doi: 10.1007/s00210-007-0168-4. Epub 2007 Jun 12. PMID 17563882
- [Result] Lu J, Yang X, Zhang J, Huang Y. The efficacy of dexmedetomidine for the prevention of catheter-related bladder discomfort: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Dec 30;100(52):e28217. doi: 10.1097/MD.0000000000028217. PMID 34967355
- [Result] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Result] Lu Y, Li Q, Wang Y, Zhou Z, Zhang D, Bao Y, Wu J, Cui Y. Meta-Analysis of the Efficacy and Safety of Ketamine on Postoperative Catheter-Related Bladder Discomfort. Front Pharmacol. 2022 Jun 27;13:816995. doi: 10.3389/fphar.2022.816995. eCollection 2022. PMID 35833034
- [Result] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Result] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Result] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Result] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Result] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Result] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Result] Akca B, Aydogan-Eren E, Canbay O, Karagoz AH, Uzumcugil F, Ankay-Yilbas A, Celebi N. Comparison of efficacy of prophylactic ketamine and dexmedetomidine on postoperative bladder catheter-related discomfort. Saudi Med J. 2016 Jan;37(1):55-9. doi: 10.15537/smj.2016.1.14122. PMID 26739975
- [Result] Agarwal A, Gupta D, Kumar M, Dhiraaj S, Tandon M, Singh PK. Ketamine for treatment of catheter related bladder discomfort: a prospective, randomized, placebo controlled and double blind study. Br J Anaesth. 2006 May;96(5):587-9. doi: 10.1093/bja/ael048. Epub 2006 Mar 10. PMID 16531445
- [Result] Agarwal A, Raza M, Singhal V, Dhiraaj S, Kapoor R, Srivastava A, Gupta D, Singh PK, Pandey CK, Singh U. The efficacy of tolterodine for prevention of catheter-related bladder discomfort: a prospective, randomized, placebo-controlled, double-blind study. Anesth Analg. 2005 Oct;101(4):1065-1067. doi: 10.1213/01.ane.0000167775.46192.e9. PMID 16192522
- [Result] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162